CLINICAL TRIAL: NCT03793842
Title: Use of Electrical Impedance Tomography for Optimization of Positive End-Expiratory Pressure in Acute Respiratory Distress Syndrome
Brief Title: Electrical Impedance Tomography for Optimization of Positive End-Expiratory Pressure: Acute Respiratory Distress Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Robert C. Hyzy, MD, Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HUM00148126
Record Dates: First submitted 2019-01-03; First posted 2019-01-04 (Actual); Results first posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-09

CONDITIONS: Acute Respiratory Distress Syndrome; ARDS
Keywords: Electrical Impedance Tomography; Ventilator; Lung; Respiration
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Aspiration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Usual care then PEEP titration by Electrical Impedance Tomography (EIT) (Experimental): Patients in the usual care first group will continue to receive mechanical ventilation according to the University of Michigan Acute Respiratory Distress Syndrome (ARDS) protocol high-PEEP arm
  Interventions: Other: Usual care; Device: PEEP titration by EIT
- PEEP titration by EIT then usual care (Experimental): Patients in the high PEEP titration by EIT first will have receive ventilation with a PEEP determined by EIT titration procedure.
  Interventions: Other: Usual care; Device: PEEP titration by EIT

INTERVENTIONS:
Other: Usual care — Intervention is the standard basic lung protective ventilation strategy used at the University Hospital Respiratory Care at Michigan Medicine.
Device: PEEP titration by EIT — PEEP Titration procedure involves two phases: a recruitment phase followed by a gradual reduction in the end-expiratory pressure phase (Decremental PEEP).
  Other Names: Drager PulmoVista 500 EIT System

SUMMARY:
Doctors follow a standard ventilator management strategy when making adjustments to the breathing machine to optimize the amount of oxygen into the lungs. The purpose of this study is to assess whether the EIT (electrical impedance tomography) device can be an additional useful tool for ventilator management and identifying the ideal positive end-expiratory pressure (PEEP).

ELIGIBILITY:
Inclusion Criteria:

* Endotracheal ventilation for < 1 week (168 hours)
* Presence of all of the following conditions for < 48 hours i. Partial pressure of oxygen to percentage of inspired oxygen (PaO2/FiO2) < 150 with PEEP > 5 cm water for > 30 min.

ii. bilateral opacities not fully explained by effusions, lobar/lung collapse, or nodules iii. respiratory failure not fully explained by cardiac failure or fluid overload

-All criteria listed in (3) developed within 1 week of a known clinical insult or new or worsening respiratory symptoms

Exclusion Criteria:

* Lack of informed consent
* Known pregnancy
* Extracorporeal membrane oxygenation (ECMO) use
* Severe chronic respiratory disease requiring home oxygen therapy or ventilation
* Calculated BMI of greater than 50

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hyzy, MD, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jimenez JV, Munroe E, Weirauch AJ, Fiorino K, Culter CA, Nelson K, Labaki WW, Choi PJ, Co I, Standiford TJ, Prescott HC, Hyzy RC. Electric impedance tomography-guided PEEP titration reduces mechanical power in ARDS: a randomized crossover pilot trial. Crit Care. 2023 Jan 17;27(1):21. doi: 10.1186/s13054-023-04315-x. PMID 36650593

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care Then Positive End-Expiratory Pressure (PEEP) Titration by EIT: Patients in the usual care first group will continue to receive mechanical ventilation according to the University of Michigan Acute Respiratory Distress Syndrome (ARDS) protocol high-PEEP arm.
  Usual care: Intervention is the standard basic lung protective ventilation strategy used at the University Hospital Respiratory Care at Michigan Medicine.
  PEEP titration by Electrical Impedance Tomography (EIT): PEEP Titration procedure involves two phases: a recruitment phase followed by a gradual reduction in the end-expiratory pressure phase (Decremental PEEP).
- Positive End-Expiratory Pressure (PEEP) Titration by EIT Then Usual Care: Patients in the high PEEP titration by Electrical Impedance Tomography (EIT) first will have receive ventilation with a PEEP determined by EIT titration procedure.
  Usual care: Intervention is the standard basic lung protective ventilation strategy used at the University Hospital Respiratory Care at Michigan Medicine.
  PEEP titration by EIT: PEEP Titration procedure involves two phases: a recruitment phase followed by a gradual reduction in the end-expiratory pressure phase (Decremental PEEP).
Period: Randomization-Intervention 1 (~6 Hrs)
Arm/Group | Usual Care Then Positive End-Expiratory Pressure (PEEP) Titration by EIT | Positive End-Expiratory Pressure (PEEP) Titration by EIT Then Usual Care
Started (Randomized) | 8 | 8
Intervention 1 Started | 6 | 6
Completed | 6 | 6
Not Completed | 2 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Prone positioning after baseline data collection | 2 | 1
Period: Intervention 2 (14-18 Hours)
Arm/Group | Usual Care Then Positive End-Expiratory Pressure (PEEP) Titration by EIT | Positive End-Expiratory Pressure (PEEP) Titration by EIT Then Usual Care
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 16 participants were randomized, 8 to each arm. 1 participant was removed because of physician's decision, while 3 were removed because of prone positioning. The 4 excluded participants are represented in the Excluded arm.
Groups:
- Usual Care Then PEEP Titration by EIT: Patients in the usual care first group will continue to receive mechanical ventilation according to the University of Michigan ARDS protocol high-PEEP arm
  Usual care: Intervention is the standard basic lung protective ventilation strategy used at the University Hospital Respiratory Care at Michigan Medicine.
  PEEP titration by EIT: PEEP Titration procedure involves two phases: a recruitment phase followed by a gradual reduction in the end-expiratory pressure phase (Decremental PEEP).
- Excluded: Patients in this arm were excluded per protocol.
- Total: Total of all reporting groups
Arm/Group | Usual Care Then PEEP Titration by EIT | PEEP Titration by EIT Then Usual Care | Excluded | Total
Number analyzed (Participants) | 6 | 6 | 4 | 16
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59.5 [46 to 67] | 62 [50 to 72] | 67 [59 to 75] | 60.5 [47 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3 | 6
  Male | 4 | 5 | 1 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 5 | 6 | 3 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 6 | 3 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Mechanical Power
Description: Mechanical power (MP) is the energy imparted to the lung from the mechanical ventilator. It is calculated as listed below, where respiratory rate = RR, tidal volume = TV, Ppeak = peak airway pressure, Pplat = plateau airway pressure and PEEP = positive end-expiratory pressure. Mechanical power determined for the difference between Treatment 1 and Treatment 2. Values shown represent data gathered at the end of the designated assignment listed below, regardless of whether that assignment was Treatment 1 or Treatment 2.
  MP = 0.098 X RR X TV (Ppeak-[Pplat-PEEP/2])
Time Frame: Participants received Treatment 1 (either Usual Care or PEEP EIT) for approximately 6 hours after randomization and then received Treatment 2 for an additional 14-18 hours following crossover. Measurement was done at end of treatment.
Population: 3 participants in whom prone ventilation was initiated were excluded. 1 additional participant was excluded due to physician withdrawal from the trial. The remaining participants received invasive mechanical ventilation in the supine position for the duration of the protocol.
Measure: Mean (Standard Deviation); unit: J/min
Groups:
- PEEP: PEEP titration by EIT: PEEP Titration procedure involves two phases: a recruitment phase followed by a gradual reduction in the end-expiratory pressure phase (Decremental PEEP).
Arm/Group | PEEP | Usual Care
Number analyzed (Participants) | 12 | 12
J/min | 1.87 (1.61) | -2.50 (3.7)
Statistical Analysis 1: Comparison: PEEP vs Usual Care; Test type: Equivalence — Equivalence margin 1 J/min; p = .002, t-test, 2 sided

2. Secondary Outcome: Change in Lung Inflammation as Measured by Physiologic Parameter: Partial Pressure of Arterial Oxygen/Fraction of Inspired Oxygen (P/F Ratio)
Description: P/F ratio is a measurement of oxygenation and, where arterial oxygen in mmHg is PaO2 and percentage of inspired oxygen is FiO2. It calculated as: PaO2/FiO2. P/F ratio determined for the difference between Intervention 1 and Intervention 2
Time Frame: Participants received Treatment 1 (either Usual Care or PEEP EIT) for approximately 6 hours after randomization and then received Treatment 2 for an additional 14-18 hours following crossover. Measurement was done at baseline and end of treatment.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | PEEP | Usual Care
Number analyzed (Participants) | 12 | 12
ratio | 25.14 (27.11) | -0.89 (60.05)
Statistical Analysis 1: Comparison: PEEP vs Usual Care; Test type: Superiority; p = 0.2, t-test, 2 sided

3. Secondary Outcome: Change in Lung Inflammation as Measured by Physiologic Parameter: Plateau Pressure
Description: Plateau pressure is a measurement of lung compliance and is the airway pressure obtained during a brief inspiratory hold after delivering a tidal volume breath during invasive mechanical ventilation. Plateau pressure determined for the difference between Intervention 1 and Intervention 2
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | PEEP | Usual Care
Number analyzed (Participants) | 12 | 12
cm H2O | 2.06 (1.88) | -2.48 (3.22)
Statistical Analysis 1: Comparison: Usual Care; Test type: Equivalence — Equivalence margin 1 cm H20; p = 0.006, t-test, 2 sided; Mean Difference (Net) = 0.05

4. Secondary Outcome: Lung Inflammation as Measured by Physiologic Parameter: Driving Pressure
Description: Driving pressure is the force of airway push into the lung while receiving invasive mechanical ventilation and is calculated as Plateau pressure - Positive end-expiratory pressure. Driving pressure determined for the difference between Intervention 1 and Intervention 2
Time Frame: as for outcome 1
Population: ARDS patients
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | PEEP | Usual Care
Number analyzed (Participants) | 12 | 12
cm H2O | 1.34 (1.31) | -1.58 (2.32)
Statistical Analysis 1: Comparison: PEEP vs Usual Care; Test type: Superiority; p = 0.003, t-test, 2 sided

5. Secondary Outcome: Change in Lung Inflammation as Measured by Physiologic Parameter: Static Compliance
Description: Static lung compliance is a measurement of lung stiffness due to disease, with a lower compliance representing stiffer lungs. It is calculated as: Tidal volume / (Plateau pressure - PEEP). Static compliance determined for the difference between Intervention 1 and Intervention 2
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: ml/cm H2O
Arm/Group | PEEP | Usual Care
Number analyzed (Participants) | 12 | 12
ml/cm H2O | 3.24 (9.85) | -4.6 (5.26)
Statistical Analysis 1: Comparison: PEEP vs Usual Care; Test type: Superiority; p = 0.008, t-test, 2 sided

6. Secondary Outcome: Partial Pressure of Arterial Oxygen (PaO2)
Description: PaO2 is the partial pressure of arterial oxygen measured in mmHg. PaO2 determined for the difference between Intervention 1 and Intervention 2.
Time Frame: as for outcome 1
Population: No PaO2 data was obtained or recorded as such. Physicians directly calculated PaO2/FiO2 data shown above in Outcome Measure 2.
Arm/Group | PEEP | Usual Care
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Dynamic Compliance (Cdyn)
Description: Dynamic compliance is a measurement of the resistance of the lungs and airways to gas installation from the mechanical ventilator and is measured as Peak airway pressure / Plateau airway pressure - PEEP). Dynamic compliance determined for the difference between Intervention 1 and Intervention 2.
Time Frame: as for outcome 1
Population: Dynamic compliance was not recorded due to the attempt of investigative personnel to limit time exposure to Coronavirus disease 19 (COVID-19) in most study participants.
Arm/Group | PEEP | Usual Care
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Compliance Over the Last 20% of Inspiration (C20/Dyn)
Description: C20 is the compliance that results when only the upper 20% of the applied pressure range is taken into account. The C20/Dyn ratio appears to effectively quantitate evidence of lung over distention during mechanical ventilation. This is a unit-less measure as both numerator and denominator are measured in cm water. C20/dyn determined for the difference between Intervention 1 and Intervention 2.
Time Frame: as for outcome 2
Population: C20/Dyn was not recorded due to the attempt of investigative personnel to limit time exposure to COVID-19 in most study participants.
Arm/Group | PEEP | Usual Care
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Ultrasound Surrogates of Lung Aeration
Description: Lung ultrasound inflation scores are calculated by summing regional scores (0-3 points), with higher scores indicating worse condition of the lung. Scores were obtained in six regions of each lung (i.e., up and down anterior, medial, and posterior chest wall). This is a unit-less measure. Ultrasound lung surrogates of lung inflation determined for the difference between Intervention 1 and Intervention 2.
Time Frame: as for outcome 1
Population: Lung ultrasound was not recorded due to the attempt of investigative personnel to limit time exposure to COVID-19 in most study participants.
Arm/Group | PEEP | Usual Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Usual Care | PEEP
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-16): https://cdn.clinicaltrials.gov/large-docs/42/NCT03793842/Prot_SAP_000.pdf